CLINICAL TRIAL: NCT00000750
Title: A Phase III Study to Evaluate the Safety, Tolerance, and Efficacy of Early Treatment With Zidovudine (AZT) in Asymptomatic Infants With HIV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 182; 11157 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
Primary: To determine the efficacy of early treatment with zidovudine (AZT) in HIV-infected asymptomatic infants. To determine the safety and tolerance of AZT in this patient population.

Secondary: To compare the virologic and immunologic parameters between the treatment groups. To determine the efficacy of AZT as an early treatment to prevent development of CD4+ cell depletion in HIV-infected asymptomatic infants.

AZT is currently indicated for primary treatment in children with HIV-associated signs and symptoms and for those with significant immunodeficiency. This study will attempt to determine whether early treatment with AZT prevents the development of symptoms in HIV-infected infants who are asymptomatic.

DETAILED DESCRIPTION:
AZT is currently indicated for primary treatment in children with HIV-associated signs and symptoms and for those with significant immunodeficiency. This study will attempt to determine whether early treatment with AZT prevents the development of symptoms in HIV-infected infants who are asymptomatic.

Patients are randomized to receive oral AZT (at age-adjusted doses) or placebo. Patients are evaluated at weeks 2 and 4 and every 4 weeks thereafter; those who reach a study endpoint will have their treatment unblinded to allow the clinician to determine which treatment regimen the patient should then receive. Patients who meet the criteria for changes to open-label AZT will be given the appropriate age-adjusted dose without unblinding the original randomization assignment. Patients who complete or discontinue treatment are followed every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4 count >= 2000 cells/mm3 AND >= 30 percent of total lymphocytes.
* No signs or symptoms of HIV infection (other than lymphadenopathy, mild hepatomegaly, hypergammaglobulinemia, or splenomegaly, which is permitted).
* Consent of parent or guardian.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Serious acute infection requiring parenteral therapy at time of entry.
* One or more serious, proven bacterial infections including any of the following:
* septicemia; pneumonia; meningitis; bone or joint infection; or abscess of an internal organ or body cavity (excluding otitis media or superficial skin or mucosal abscesses) that are caused by Haemophilus, Streptococcus (including pneumococcus), or other pyogenic bacteria.
* Clinical neurologic/neuropsychologic deficits, or a head circumference less than the fifth percentile.

Concurrent Medication:

Excluded:

* Any agent with known antiretroviral activity.
* Acetaminophen, ibuprofen, or aspirin for more than 72 hours continuously.

Prior Medication:

Excluded:

* More than 7 weeks of prior antiretroviral or immunomodulator therapy post-natally.

Recommended:

* PCP prophylaxis.
* Immunizations according to current recommendations.

Ages: 1 Day to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E Connor, Study Chair; G McSherry, Study Chair
Locations (42):
- United States (41):
  - Univ of Alabama at Birmingham Schl of Med / Pediatrics, Birmingham, Alabama
  - Kaiser Permanente / UCLA Med Ctr, Downey, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Children's Hosp of Denver, Denver, Colorado
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Yale Univ Med School, New Haven, Connecticut
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Miami (Pediatric), Miami, Florida
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - King's County Hosp Ctr / Pediatrics, Brooklyn, New York
  - Children's Hosp Pact Prog / Children's Hosp of Buffalo, Buffalo, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Lincoln Hosp Ctr, The Bronx, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Westchester Hosp, Valhalla, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Columbus Children's Hosp, Columbus, Ohio
  - Med Univ of South Carolina, Charleston, South Carolina
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
- San Juan City Hosp, San Juan, Puerto Rico